CLINICAL TRIAL: NCT06056765
Title: Effect of ESWT Versus Exercise Treatment for Thumb Carpometacarpal Osteoarthritis: a Randomized Trial.
Brief Title: Extracorporeal Shock Waves Therapy (ESWT) vs Exercise in Thumb Osteoarthritis
Acronym: SWEX-TO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWEX-TO
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Thumb Osteoarthritis; Hand Injuries
Keywords: shock waves; exercise; conservative treatment; hand
MeSH Terms: conditions — Hand Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT group (Experimental): The therapy will be applied using a focused shock wave device ("Minilith", Storz, Swiss) at the pulley of the first extensor channel under ultrasound guidance. Shock wave therapy will be performed with the patient's hand in intermediate between pronation and supination and will be administered once a week, for 3 sessions. For each treatment session, 2000 pulses will be applied with an energy flux density of 0.09 mJ/mm2 (between 0.05 and 0.12 mJ/mm2) and a frequency of 4 pulses per second (4 Hz). Gel will be used between the probe and the skin during applications to ensure conductivity. No local anesthetic will be used. Patients in both groups will be instructed to use a brace during the day for 4 weeks following recruitment.
  Interventions: Device: "Minilith", Storz, Swiss
- Exercise group (No Intervention): Patients will perform exercises for 4 weeks following recruitment. Patients in this group will be taught home exercises to improve the dynamic stability of the thumb metacarpal trapezius joint. The patient is instructed to perform a flexion of the trapeziometacarpal. If the individual is able to complete 10 repetitions with good technique, resistance will be added manually or with rubber bands. If this exercise is painful, they are asked to return to active movement only. Patients in both groups will be instructed to use a brace during the day for 4 weeks following recruitment.

INTERVENTIONS:
Device: "Minilith", Storz, Swiss — shock waves
  Other Names: Extracorporeal Shock Waves Therapy; ESWT
  Arms: ESWT group

SUMMARY:
Osteoarthritis (OA) is a chronic joint disease with a high prevalence and a negative impact on the quality of life and a high economic burden. The most common form of OA is that involving the hands, which affects females three times more often. OA of the base of the first finger is present in 21% of the population over 40 years of age and is more frequently related to pain and disability than OA of the interphalangeal joint. In addition to pain, it can cause deformity, stiffness, reduced mobility and strength, resulting in difficulty performing common activities such as opening vessels, carrying weights and writing.

OA of the base of the first toe is mainly treated with conservative modalities, while surgical treatment will be reserved for those whose debilitating symptoms persist despite adequate conservative management. Surgical management, however, is associated with a number of complications, including tendon rupture, sensory changes, and wound infection.

Although a number of conservative therapies have proven effective for the management of hand OA, there are few high-quality clinical studies in the literature to date.

DETAILED DESCRIPTION:
The review of the literature has shown that in thumb carpometacarpal osteoarthritis the use of braces leads to a reduction in pain, particularly in the long term, based on data from two studies. Additionally, hand exercises could improve grip strength and hand function.

Regarding pharmacological management, insufficient data are available to support the effectiveness of intra-articular therapy with corticosteroids or hyaluronic acid and their use is not recommended by the American College of Rheumatology guidelines (ACR) of 2012 . On the other hand, nonsteroidal anti-inflammatory drugs (NSAIDs) are recommended to relieve pain associated with first toe base OA, and topical formulations are recommended over oral NSAIDs in more recent guidelines, due to a profile of superior security. However, their effect on function is minimal and transient (no more effective than placebo after 2 weeks).

The combination of non-pharmacological and pharmacological modalities in the management of hand OA is recommended by the European League Against Rheumatism (EULAR) guidelines and is frequently used in clinical practice. Despite this, direct evidence of the effectiveness of this strategy is lacking. There have been some studies evaluating combined treatment, although they have generally not been specific to OA of the base of the first toe. Furthermore, the combinations studied usually included exclusively nonpharmacological modalities, and to date no strategy has been found to be highly effective for improving pain and function for first toe base OA.

Determining an evidence-based treatment approach with a clinically significant effect on clinical outcomes would provide healthcare providers with a basis for decision making for the treatment of patients with thumb carpometacarpal osteoarthritis. This strategy does not yet exist, and decisions about the best combination of interventions are generally based on personal experience and the personal opinion of healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* arthrosis of the trapezoid-metacarpal with stage 1 or 2 of the Eaton-Littler radiographic classification and pain (recent radiograph within 6 months previously);
* clinical picture that has been occurring for at least 6 months;
* pain scored with VAS scale at least 4/10.

Exclusion Criteria:

* rheumatoid arthritis or outcomes of trauma in the affected area,
* contra-indications to treatment with shock waves (neoplasia, pregnancy, thrombocytopenia, epilepsy, uncompensated heart disease or arrhythmia, pacemaker, local infections),
* corticosteroid infiltration or physical therapy in the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
recovery of pain | change between baseline to 1 month
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
recovery of pain | change between baseline to 3 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
recovery of pain | change between baseline to 6 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
recovery of pain | change between baseline to 12 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
functional recovery | change between baseline to 1 month
  The Functional Index of Hand Osteoarthritis (FIHOA) measures the effect of hand problems on function in terms of pain and disability.The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 30; the higher the score, the more limitation/pain/disability is present.
functional recovery | change between baseline to 3 months
  The Functional Index of Hand Osteoarthritis (FIHOA) measures the effect of hand foot problems on function in terms of pain and disability.The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 30; the higher the score, the more limitation/pain/disability is present.
functional recovery | change between baseline to 6 months
  The Functional Index of Hand Osteoarthritis (FIHOA) measures the effect of hand problems on function in terms of pain and disability.The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 30; the higher the score, the more limitation/pain/disability is present.
functional recovery | change between baseline to 12 months
  The Functional Index of Hand Osteoarthritis (FIHOA) measures the effect of hand problems on function in terms of pain and disability.The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 30; the higher the score, the more limitation/pain/disability is present.
disability recovery | change between baseline to 1 month
  The Disabilities of the Arm, Shoulder and Hand Score (QuickDash) contains 11 questions related to ability and pain in the past week. Scores range from 0 to 100; the higher the score, the greater the limitation/pain/disability.
disability recovery | change between baseline to 3 months
  The Disabilities of the Arm, Shoulder and Hand Score (QuickDash) contains 11 questions related to ability and pain in the past week. Scores range from 0 to 100; the higher the score, the greater the limitation/pain/disability.
disability recovery | change between baseline to 6 months
  The Disabilities of the Arm, Shoulder and Hand Score (QuickDash) contains 11 questions related to ability and pain in the past week. Scores range from 0 to 100; the higher the score, the greater the limitation/pain/disability.
disability recovery | change between baseline to 12 months
  The Disabilities of the Arm, Shoulder and Hand Score (QuickDash) contains 11 questions related to ability and pain in the past week. Scores range from 0 to 100; the higher the score, the greater the limitation/pain/disability.
perception of clinical improvement | change between 3 to 6 months
  Maudsley and Roles scale scores range from 0-4 points for excellent to poor
perception of clinical improvement | change between 3 to 12 months
  Maudsley and Roles scale scores range from 0-4 points for excellent to poor

CONTACTS AND LOCATIONS:
Locations (1):
- Angela Notarnicola, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lane LB, Boretz RS, Stuchin SA. Treatment of de Quervain's disease:role of conservative management. J Hand Surg Br. 2001 Jun;26(3):258-60. doi: 10.1054/jhsb.2001.0568. PMID 11386780
- [Background] Stepan JG, London DA, Boyer MI, Calfee RP. Blood glucose levels in diabetic patients following corticosteroid injections into the hand and wrist. J Hand Surg Am. 2014 Apr;39(4):706-12. doi: 10.1016/j.jhsa.2014.01.014. PMID 24679910
- [Background] Cavaleri R, Schabrun SM, Te M, Chipchase LS. Hand therapy versus corticosteroid injections in the treatment of de Quervain's disease: A systematic review and meta-analysis. J Hand Ther. 2016 Jan-Mar;29(1):3-11. doi: 10.1016/j.jht.2015.10.004. Epub 2015 Nov 6. PMID 26705671
- [Background] Brinks A, Koes BW, Volkers AC, Verhaar JA, Bierma-Zeinstra SM. Adverse effects of extra-articular corticosteroid injections: a systematic review. BMC Musculoskelet Disord. 2010 Sep 13;11:206. doi: 10.1186/1471-2474-11-206. PMID 20836867
- [Background] Peters-Veluthamaningal C, Winters JC, Groenier KH, Meyboom-DeJong B. Randomised controlled trial of local corticosteroid injections for de Quervain's tenosynovitis in general practice. BMC Musculoskelet Disord. 2009 Oct 27;10:131. doi: 10.1186/1471-2474-10-131. PMID 19860883
- [Background] Kjeken I, Smedslund G, Moe RH, Slatkowsky-Christensen B, Uhlig T, Hagen KB. Systematic review of design and effects of splints and exercise programs in hand osteoarthritis. Arthritis Care Res (Hoboken). 2011 Jun;63(6):834-48. doi: 10.1002/acr.20427. PMID 21630479
- [Background] Trellu S, Dadoun S, Berenbaum F, Fautrel B, Gossec L. Intra-articular injections in thumb osteoarthritis: A systematic review and meta-analysis of randomized controlled trials. Joint Bone Spine. 2015 Oct;82(5):315-9. doi: 10.1016/j.jbspin.2015.02.002. Epub 2015 Mar 14. PMID 25776442
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Zhang W, Doherty M, Leeb BF, Alekseeva L, Arden NK, Bijlsma JW, Dincer F, Dziedzic K, Hauselmann HJ, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Maheu E, Martin-Mola E, Pavelka K, Punzi L, Reiter S, Sautner J, Smolen J, Verbruggen G, Zimmermann-Gorska I. EULAR evidence based recommendations for the management of hand osteoarthritis: report of a Task Force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2007 Mar;66(3):377-88. doi: 10.1136/ard.2006.062091. Epub 2006 Oct 17. PMID 17046965
- [Background] Henry KD, Rosemond C, Eckert LB. Effect of number of home exercises on compliance and performance in adults over 65 years of age. Phys Ther. 1999 Mar;79(3):270-7. PMID 10078770
- [Background] O'Brien VH, Giveans MR. Effects of a dynamic stability approach in conservative intervention of the carpometacarpal joint of the thumb: a retrospective study. J Hand Ther. 2013 Jan-Mar;26(1):44-51; quiz 52. doi: 10.1016/j.jht.2012.10.005. Epub 2012 Nov 21. PMID 23177671
- [Background] Mobargha N, Esplugas M, Garcia-Elias M, Lluch A, Megerle K, Hagert E. The effect of individual isometric muscle loading on the alignment of the base of the thumb metacarpal: a cadaveric study. J Hand Surg Eur Vol. 2016 May;41(4):374-9. doi: 10.1177/1753193415597114. Epub 2015 Aug 6. PMID 26253421
- [Background] Pellegrini VD Jr. Osteoarthritis at the base of the thumb. Orthop Clin North Am. 1992 Jan;23(1):83-102. PMID 1729673
- [Background] Moulton MJ, Parentis MA, Kelly MJ, Jacobs C, Naidu SH, Pellegrini VD Jr. Influence of metacarpophalangeal joint position on basal joint-loading in the thumb. J Bone Joint Surg Am. 2001 May;83(5):709-16. doi: 10.2106/00004623-200105000-00009. PMID 11379740
- [Background] Pisano K, Wolfe T, Lubahn J, Cooney T. Effect of a stabilization exercise program versus standard treatment for thumb carpometacarpal osteoarthritis: A randomized trial. J Hand Ther. 2023 Jul-Sep;36(3):546-559. doi: 10.1016/j.jht.2022.03.009. Epub 2022 Jul 8. PMID 35811182